CLINICAL TRIAL: NCT02702583
Title: The Oral Cavity as a Source of Febrile Neutropenia: An Observational Study in Cancer Patients Treated With Myelosuppressive Chemotherapy
Brief Title: The Oral Cavity as a Source of Febrile Neutropenia
Acronym: ORA-FEBRIS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.A.E.M. Zecha, Phd student, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL53440.018.15
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Febrile Neutropenia; Solid Tumors; Dental Infection; Oral Infection
Keywords: Myelosuppressive Chemotherapy; Febrile Neutropenia; Solid Tumors; Dental Infection; Oral Infection
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral rinsing samples
  Saliva samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Febrile neutropenia (FN) is a clinically important adverse effect of myelosuppressive chemotherapy. If patients present with FN, attention is focussed on well-recognized sites of origin of infection: the airways, urinary tracts, and skin. However, infections can be only documented clinically in about two-third of febrile episodes, whereas a causative microbial pathogen cannot be identified in the majority (>70%) of cases.

Pre-treatment oral evaluation aimed to identify and eliminate oral/dental foci is only routinely used in patients at high risk for oral complications (i.e. head and neck cancer patients and stem cell transplantation recipients). However, any patient treated with myelosuppressive chemotherapy, be it for cure or palliation, is at risk of developing infection in and/or originating from the oral cavity. Nevertheless, in these patients dental screening is somewhat randomly employed at the oncologist's discretion.

More insight into the pre-treatment oral condition and its potential role in FN is mandatory, particularly considering the growing numbers of older patients retaining their natural dentition and the increase of dental diseases and cancer incidence with age.

In addition, oral diseases may aggravate chemotherapy-induced oral mucositis (OM). OM is associated with an inflammatory response, which together with ulcerations providing a portal of entry for bacteria, can result in FN and systemic inflammatory syndrome (SIRS) and/or sepsis. Evidence suggests that microorganisms are involved in the pathobiology of OM, but no longitudinal studies using open-end sequencing are available.

Furthermore, comparing bacteria identified in blood cultures in febrile patients with those of the oral cavity will expand the knowledge on the role of the oral cavity as a potential source of bacteremia.

The investigators expect that the results will provide a scientific base for subsequent intervention studies on the efficacy of dental screening and elimination of foci, and other interventions aimed at modifying the oral environment before and during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a solid cancer, lymphoma or multiple myeloma
* Planned treatment with myelosuppressive chemotherapy with FN risk of 10%-20% (with or without targeted therapies or hormonal therapy)
* Willing and able to give written Informed consent
* Age 18 or older
* Presence of (partial) natural dentition and/or dental implants

Exclusion Criteria:

* Patients unable to give written informed consent
* Patients <18 years
* Prior irradiation to the head and neck
* Edentulous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with myelosuppressive chemotherapy with a 10-20% estimated risk to develop febrile neutropenia.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Dutch Periodontal Screening Index | 1 day
  Score Clinical criteria for the score per sextant (note site per sextant with the highest score) 0 No pockets >3mm in depth, no calculus, no overhanging restorations and no bleeding on probing to the bottom of the pocket
  1. No pockets >3mm in depth, no calculus, no overhangs of restorations, but presence of bleeding on probing to the bottom of the pocket
  2. No pockets >3mm in depth, presence of bleeding on probing to the bottom of the pocket, and presence of calculus or overhanging restorations
  3. Presence of pathological pockets of 4-5mm without gingival recession
  4. Presence of pathological pockets of 4-5mm with gingival recession
  5. Presence of pathological pockets of 6mm or more.
  Ref:
  Van der Velden U, (2009) J Clin Periodontol. 2009 Dec;36(12):1018-24. doi: 10.1111/j.1600-051X.2009.01495.x.
  The Dutch periodontal screening index validation and its application in The Netherlands.
Caries-screening | 1 day
  1. no caries
  2. caries in enamel
  3. caries <50% in dentin
  4. caries >50% in dentin
  5. caries in rootcanal
Impacted (wisdom) teeth | 1 day
  1. not impacted
  2. partially impacted
  3. impacted
Plaque index in percentages | 1 day
  The plaque index is calculated via the amount of plaque on the mesiobuccal+buccal+distobuccal+mesiopalatinal or mesiolingual+palatinal or lingual+distopalatinal or distolingual of every tooth, given in percentages.
Radiographically (X-OPT) calculated bone loss in millimeters | 1 day
  Bone loss is measured on a X-OPT and the average bone loss is noted in millimeters.
Peri-apical radiolucency | 1 day
  Peri-apical radiolucency is diagnosed on a X-OPT or intraoral radiograph and will be noted as
  1. yes
  2. no
Radix relicta | 1 day
  The presence of radix relicta is noted as
  1. yes
  2. no

SECONDARY OUTCOMES:
NCI CTCAE V3.0 mucositis/stomatitis | 100 days
  The NCI-CTCAE v3.0 mucositis/stomatitis is noted for every patient when visiting the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: L. Smeele, Professor, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands